CLINICAL TRIAL: NCT04559906
Title: Effects of Spray and Stretch Technique Versus Sustain Pressure for the Management of Upper Trapezius Triggers
Brief Title: Spray Stretch Technique Versus Sustain Pressure for Trapezius Triggers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00686 Uzair Ahmad
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Trigger Point Pain, Myofascial; Mechanical Neck Pain
Keywords: Spray and Stretch technique; Progressive Pressure release technique; Active myofascial trigger points; Upper Trapezius Triggers
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Ethyl Chloride

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Spray and Stretch technique Conventional treatment Hot pack (10-15 min) Stretching (3 sets of 10 repetitions with 10 seconds hold) AROM exercises (3 sets of 10 repetition)
  Interventions: Other: Spray and Stretch technique (Ethyl chloride)
- Group B (Active Comparator): Sustain pressure release Conventional treatment Hot pack (10-15 min) Stretching (3 sets of 10 repetitions with 10 seconds hold) AROM exercises (3 sets of 10 repetition)
  Interventions: Other: Sustain pressure release

INTERVENTIONS:
Other: Spray and Stretch technique (Ethyl chloride) — Group A receive spray and stretch technique (Ethyl chloride) with conventional treatment.
  The upper trapezius muscle stretches on the basis of the Technique originally described by Simons. The subject is seated in a relaxed position on their homolateral hand for anchoring the distal end of the studied muscle. Initially, 3 to 5 parallel sweeps of ethyl chloride spray is applied covering the Upper trapezius muscle. Then, the muscle are positioned in a maximal but tolerable stretch and lengthened until the Physical Therapist felt the muscle tension barrier. This procedure repeated 2 or 3 times.
  Arms: Group A
Other: Sustain pressure release — Group B receive sustain pressure release with conventional treatment. Progressive pressure release are considered in two stages. The initial step is to recognize and find the trigger in upper fiber of trapezius, utilizing trigger point palpation. Trigger point felt as firm and restricted hyperirritable knots with in gut of the muscle.
  The second step is to applying pressure release ranging from eight to twelve second for each pressure, then it increases gradually for maximum of twenty seconds. The total duration of pressure is five minutes or more until the discharge is felt by the fingers.
  Arms: Group B

SUMMARY:
The aim of this research is to determine the effects of spray and stretch technique versus sustain pressure for the management of upper trapezius triggers. A randomized control trail is conducting at Khyber Teaching Hospital Peshawar and Northwest General Hospital and Research center Peshawar. The sample size is 54. The Participants divide into two groups, 27 participants in Group A (receive the spray and stretch technique) and 27 in Group B (receive sustain pressure). The study duration is 6 months. Purposive non probability sampling technique applied. Only 20 to 35 years participants with upper trapezius trigger is including in this trial. Tools use in this study are visual analogue scale (VAS), Neck Disability Index (NDI), Hospital Anxiety and Depression Scale (HADS), Goniometer, Algometer and Manual muscle strength (MMT). Data analyzed through SPSS version 25.

DETAILED DESCRIPTION:
Myofascial Trigger Point (MTrP) is a hyperirritable spot in the taut bands of the skeletal muscles' fascia which is palpable and tender, on direct compression can produce referred pain in its reference zone, local tenderness and elicit a local twitch response. MTrP can be identified as either active or latent. According to Simons et al. that active and latent trigger points are associated with tenderness, muscle dysfunction, muscle weakness and restricted muscle length. An active MTrP causes spontaneous pain complaint in surrounding tissue and generally in its pain reference zone while latent MTrP physically exist but doesn't associate with spontaneous pain complaint. However, by direct compression latent MTrP can cause local pain on the site of taut band. Myofascial trigger points (MTrP) are considered one of the most common cause of musculoskeletal pain. Active MTrP are considered to be more prevalent in upper fibers of trapezius muscle (45% in right upper trapezius and 25% in left upper trapezius and cause neck pain and shoulder discomfort. Predisposing Factors associated to MTrP can be either mechanical stress (such as overuse of muscles, repetitive strain injury, work related mechanical disorder, awkward posture and degenerative condition) or metabolic stress( such as hypo metabolic state and vitamin deficiency).According to integrated hypothesis presented by Simon, MTrP is believed to develop after a local injury either repetitive micro trauma or gross trauma to the muscle fibers. The diagnostic criteria of MTrP used by recent studies which is presented by Simons et al. is based on palpation of muscle. A well-trained clinician palpates the muscle to localize the active MTrP. During physical examination, a hyper sensitive spot within taut bands of muscle fibers, Palpation of recognized spot results in referred pain within reference zone, palpation of recognized spot elicits a jump sign (defensive movement), palpation may result in local twitch response defined as visible contraction of muscle. There are varieties of physiotherapy interventions for the management of MTrP which maybe invasive and non-invasive such as dry needling, anesthetic injections, spray and stretch, ischemic compression and muscle energy techniques. A very limited evidence found on effects of spray and stretch technique versus sustain pressure for the Management of upper trapezius trigger points with flaws in methodology design. To fill the gap, this study is formulated to determine the effects of spray and stretch technique vs sustain pressure for the management of upper trapezius MTrP. Study will find out most effective treatment for management of upper trapezius and would contribute to educate and treat the patient with most simple and effective treatment approach.

Literature review A systematic and evidence-based search of relevant literature were performed by utilizing PubMed and Google Scholar as search engines.

A study conducted in 2017 regarding spray and stretch technique versus progressive pressure release on treatment of myofascial pain trigger point reported that spray and stretch technique was more effective in increasing functional activities while progressive pressure release was more effective in decreasing pain

Another study in 2017 regarding Immediate effect of spray and stretch on trapezitis demonstrated that spray and stretch technique is effective in terms to increases range of motion and increase pain pressure threshold on acute trapezitis.

A study in 2017 found that the number of active MTrP was positively associated with the physical burden of headache and trait anxiety.

Study in 2013 concluded that Vapocoolant spray may be more effective than ice as an analgesic for IV insertion. Subjects were more satisfied with vapocoolant spray.

Another study in 2014 investigated that spray and stretch had a short-term (<6h) effect in reducing post needling soreness of a latent MTrP and Pressure pain threshold did not significantly change after spray and stretch.

Study in 2018 reported that ischemic compression and progressive sustained pressure both have significant effect on improving the pain of patients with chronic musculoskeletal pain pathologies.

ELIGIBILITY:
Inclusion Criteria:

* At least one active myofascial trigger point in upper trapezius muscle.
* Painful limitation of neck lateral flexion range to opposite side of affected muscle.

Exclusion Criteria:

* Participants with pain pattern which is similar to pain of trigger point due to any other reason not related myofascial trigger points.
* Any trauma to cervical spine (whiplash injury) or any cervical spine surgery.
* Cervical myeloma, complex regional pain syndrome, thoracic outlet syndrome.
* Cervical radiculopathy

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 2 weeks
  Changes from base line Northwick disability index was developed first in Northwick Park hospital, England. It was designed to measure the neck pain and disability over time. It consists of 10, five parts sections. At the end, score is calculated by dividing the obtained score by total (50) multiplied by 100.
Pressure Pain Threshold (PPT) | 2 weeks
  Changes from the Baseline Pressure Pain Threshold (PPT) will taken with the help of Algometer

SECONDARY OUTCOMES:
Visual Analogue scale(VAS) | 2 weeks
  Changes from base Line Visual Analogue scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain
Range Of Motion of cervical | 2 weeks
  Changes from the Baseline range of Motion of cervical spine will take with the Help of Goniometer
The Hospital Anxiety and Depression Scale (HADS) | 2 weeks
  HADS is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. The HADS is a fourteen-item scale. Seven of the items relate to anxiety and seven relate to depression.The "0-7" score indicates normal condition,"8-10" score indicates boarderline case and "11-21" score indicates the abnormal case.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Saira Waqqar, PP-DPT,MHPE, Principal Investigator — Riphah International University
Locations (1):
- Northwest General hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amin D. SPRAY STRETCH TECHNIQUE VERSUS PROGRESSIVE PRESSURE RELEASE ON TRATMENT OF MYOFACIAL PAIN TRIGGER POINT: RANDOMIZED CONTROLLED TRIAL. International Journal of Physiotherapy and Research. 2017;5:2101-7
- [Background] Bulbuli D. Immediate Effect of Spray and Stretch Technique on Trapezits: An Experimental Study. Journal of Medical Science And clinical Research. 2017;05:20591-6
- [Background] Palacios-Cena M, Castaldo M, Wang K, Catena A, Torelli P, Arendt-Nielsen L, Fernandez-de-Las-Penas C. Relationship of active trigger points with related disability and anxiety in people with tension-type headache. Medicine (Baltimore). 2017 Mar;96(13):e6548. doi: 10.1097/MD.0000000000006548. PMID 28353618
- [Background] Waterhouse MR, Liu DR, Wang VJ. Cryotherapeutic topical analgesics for pediatric intravenous catheter placement: ice versus vapocoolant spray. Pediatr Emerg Care. 2013 Jan;29(1):8-12. doi: 10.1097/PEC.0b013e31827b214b. PMID 23283254
- [Background] Martin-Pintado Zugasti A, Rodriguez-Fernandez AL, Garcia-Muro F, Lopez-Lopez A, Mayoral O, Mesa-Jimenez J, Fernandez-Carnero J. Effects of spray and stretch on postneedling soreness and sensitivity after dry needling of a latent myofascial trigger point. Arch Phys Med Rehabil. 2014 Oct;95(10):1925-1932.e1. doi: 10.1016/j.apmr.2014.05.021. Epub 2014 Jun 10. PMID 24928191
- [Background] Sharifullah M, Sajjad A, Mubeen A, Tariq I, Khan A, Darain H. COMPARISON OF SUSTAINED PRESSURE VS ISCHEMIC COMPRESSION ON TRIGGER POINTS IN CHRONIC MYOFACIAL PAIN MANAGEMENT. 2018